CLINICAL TRIAL: NCT02253290
Title: Neuropsychological and Psychosocial Follow up of Children and Adolescents With Neuromuscular Disease
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S57182
Record Dates: First submitted 2014-09-18; First posted 2014-10-01 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Neuromuscular Diseases
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 18 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neuromuscular disease: Children and adolescents with Neuromuscular disease children according to neuromuscular convention UZL

SUMMARY:
This project is a retrospective and prospective investigation of neuropsychological and psychosocial development of children with a neuromuscular disease.

DETAILED DESCRIPTION:
This project is a retrospective and prospective investigation of neuropsychological and psychosocial development of children with a neuromuscular disease. Children and adolescents in UZ Leuven will be evaluated according to a psychosocial and neuropsychological protocol including different psychological tests and patient questionaires.

ELIGIBILITY:
Inclusion criteria

* children and adolescents (0-18 years)
* diagnosis of neuromuscular disease

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children and adolescents with neuromuscular disease
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-12 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological profile (questionnaires, neuropsychological testing) of children with myotonic dystonia type 1 | one year
  Compare the outcome of the questionnaires, IQ test and other neuropsychological test to a normal population

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Goemans, MD, PhD, Principal Investigator — UZ Leuven; Liesbeth De Waele, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium